CLINICAL TRIAL: NCT06470347
Title: A Real-World Study of Pyrrolitinib Maleate Tablets for HER-2-Positive Early or Locally Advanced Breast Cancer After Adjuvant Trastuzumab Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, LV Junyuan, Doctor of Medicine, Principal Investigator, Zunyi Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZMU-BRCA-1
Record Dates: First submitted 2024-03-24; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: HER-2 Positive Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrrolitinib (Experimental): Subjects will receive 52 weeks (approximately 1 year) of continuous oral administration of piretinib, 400 mg administered once daily, within 30 minutes of breakfast.
  Interventions: Drug: A Real-World Study of Pyrrolitinib Maleate Tablets for HER-2-Positive Early or Locally Advanced Breast Cancer After Adjuvant Trastuzumab Therapy

INTERVENTIONS:
Drug: A Real-World Study of Pyrrolitinib Maleate Tablets for HER-2-Positive Early or Locally Advanced Breast Cancer After Adjuvant Trastuzumab Therapy — During treatment, subjects were given 400 mg pyrrotinib once daily, within 30 minutes after breakfast.
  Other Names: pyrrolitinib

SUMMARY:
Purpose of the Study:

Primary Study Objective:

To evaluate the efficacy of pyrrolitinib maleate tablets in the treatment of HER-2-positive early or locally advanced breast cancer after adjuvant therapy with trastuzumab

Secondary Research Objectives:

To evaluate the safety of pyrrolitinib maleate tablets in the treatment of HER-2 positive early or locally advanced breast cancer after trastuzumab adjuvant therapy

Study Endpoints Primary Study Endpoint:

Invasive disease free survival (iDFS)

Secondary Study Endpoints:

1. overall survival (OS);
2. disease-free survival (DFS);
3. distant metastasis free survival (DDFS);
4. safety Study Population: Patients with early or locally advanced HER-2 positive breast cancer with clinical stage 0-III who have received prior neoadjuvant or adjuvant therapy. where the neoadjuvant and/or adjuvant treatment phase has been completed at least ≥24 weeks (8 dosing cycles) of trastuzumab therapy and the time interval between the end of the last course of trastuzumab therapy and entry into the study must be ≤1 year Study Design: Single-arm, multicenter, interventional study Administration Pyrrolitinib: The recommended dose of this product is 400 mg orally once daily within 30 minutes after breakfast for 52 weeks (approximately one year).

Dose adjustments may be made in accordance with this protocol, taking into account adverse reactions in subjects. Each consecutive suspension of piretinib during the course of the study should not exceed 14 days, prophylactic use of medications for the treatment of diarrhea is permitted during the course of treatment, multiple suspensions of study medication due to adverse events are permitted, and doses of piretinib that are missed for any reason will not be made up.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years;
* Invasive breast cancer with clinical stage 0-III and treated surgically;
* Histopathologically confirmed HER-2 positivity: immunohistochemistry (IHC) result of 3+ or in situ hybridization (ISH) result of HER-2 gene amplification (HER-2/CEP17 ≥ 2.0 or average HER-2 copy number/cell ≥ 6);
* Have undergone radical mastectomy or breast-conserving surgery for breast cancer, with no cancer left in the body and no recurrence of metastatic disease after surgery:

  1. Pathologic test confirms that there is no residual invasive cancer at the margins and no residual ductal carcinoma in situ;
  2. Patients who have not received neoadjuvant therapy should have negative surgical margins, and there is no requirement for the presence of lymph node metastasis (including the presence of lymph node micrometastasis) suggested by postoperative pathological tests;
  3. Patients receiving neoadjuvant therapy are not allowed to have postoperative pathologic evidence of invasive carcinoma in the breast or axillary lymph nodes;
* Previous trastuzumab anti-HER-2 therapy: completion of ≥24 weeks (8 dosing cycles) of trastuzumab in the neoadjuvant and/or adjuvant phases; the interval between the end of the last course of trastuzumab therapy and entry into the study must be ≤1 year.
* Known hormone receptor status (ER/PR);
* ECOG score of 0-1;

Normal function of major organs:

1. Blood count:

   Neutrophils (ANC) ≥ 1.5 x 109/L; Platelet count (PLT) ≥90×109/L; Hemoglobin (Hb) ≥90 g/L;
2. Blood biochemistry:

   Total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 × ULN; Alkaline phosphatase ≤ 2.5 x ULN; Urea or urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN;
3. Cardiac ultrasound:

   Left ventricular ejection fraction (LVEF) ≥55%;
4. 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) < 470 msec.

   * For female patients who are not menopausal or surgically sterilized: consent to abstinence or use of an effective non-hormonal pharmacologic method of contraception for the duration of treatment and for 8 weeks after the last dose of study treatment;
   * Benefit in the opinion of the investigator;
   * Voluntarily participate in the study by signing an informed consent form.

Exclusion Criteria:

* Confirmed local/regional recurrence/metastasis at enrollment;
* Prior anti-HER-2 therapy with pyrrolitinib, lenatinib, lapatinib and other tyrosine kinase inhibitors;
* History of gastrointestinal disease with diarrhea as the primary symptom;
* Psychiatric illness or psychotropic substance abuse that prevents cooperation;
* Female patients who are pregnant or breastfeeding;
* Those who, in the opinion of the investigator, are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival | 18 months Max

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Slamon DJ, Clark GM, Wong SG, Levin WJ, Ullrich A, McGuire WL. Human breast cancer: correlation of relapse and survival with amplification of the HER-2/neu oncogene. Science. 1987 Jan 9;235(4785):177-82. doi: 10.1126/science.3798106.
- [Background] Paik S, Hazan R, Fisher ER, Sass RE, Fisher B, Redmond C, Schlessinger J, Lippman ME, King CR. Pathologic findings from the National Surgical Adjuvant Breast and Bowel Project: prognostic significance of erbB-2 protein overexpression in primary breast cancer. J Clin Oncol. 1990 Jan;8(1):103-12. doi: 10.1200/JCO.1990.8.1.103. PMID 1967301
- [Background] Cossetti RJ, Tyldesley SK, Speers CH, Zheng Y, Gelmon KA. Comparison of breast cancer recurrence and outcome patterns between patients treated from 1986 to 1992 and from 2004 to 2008. J Clin Oncol. 2015 Jan 1;33(1):65-73. doi: 10.1200/JCO.2014.57.2461. Epub 2014 Nov 24. PMID 25422485
- [Background] Michaelson JS, Silverstein M, Sgroi D, Cheongsiatmoy JA, Taghian A, Powell S, Hughes K, Comegno A, Tanabe KK, Smith B. The effect of tumor size and lymph node status on breast carcinoma lethality. Cancer. 2003 Nov 15;98(10):2133-43. doi: 10.1002/cncr.11765. PMID 14601082
- [Background] Voduc KD, Cheang MC, Tyldesley S, Gelmon K, Nielsen TO, Kennecke H. Breast cancer subtypes and the risk of local and regional relapse. J Clin Oncol. 2010 Apr 1;28(10):1684-91. doi: 10.1200/JCO.2009.24.9284. Epub 2010 Mar 1. PMID 20194857
- [Background] Goldhirsch A, Gelber RD, Piccart-Gebhart MJ, de Azambuja E, Procter M, Suter TM, Jackisch C, Cameron D, Weber HA, Heinzmann D, Dal Lago L, McFadden E, Dowsett M, Untch M, Gianni L, Bell R, Kohne CH, Vindevoghel A, Andersson M, Brunt AM, Otero-Reyes D, Song S, Smith I, Leyland-Jones B, Baselga J; Herceptin Adjuvant (HERA) Trial Study Team. 2 years versus 1 year of adjuvant trastuzumab for HER2-positive breast cancer (HERA): an open-label, randomised controlled trial. Lancet. 2013 Sep 21;382(9897):1021-8. doi: 10.1016/S0140-6736(13)61094-6. Epub 2013 Jul 18. PMID 23871490
- [Background] Martin M, Holmes FA, Ejlertsen B, Delaloge S, Moy B, Iwata H, von Minckwitz G, Chia SKL, Mansi J, Barrios CH, Gnant M, Tomasevic Z, Denduluri N, Separovic R, Gokmen E, Bashford A, Ruiz Borrego M, Kim SB, Jakobsen EH, Ciceniene A, Inoue K, Overkamp F, Heijns JB, Armstrong AC, Link JS, Joy AA, Bryce R, Wong A, Moran S, Yao B, Xu F, Auerbach A, Buyse M, Chan A; ExteNET Study Group. Neratinib after trastuzumab-based adjuvant therapy in HER2-positive breast cancer (ExteNET): 5-year analysis of a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1688-1700. doi: 10.1016/S1470-2045(17)30717-9. Epub 2017 Nov 13. PMID 29146401
- [Background] Ma F, Li Q, Chen S, Zhu W, Fan Y, Wang J, Luo Y, Xing P, Lan B, Li M, Yi Z, Cai R, Yuan P, Zhang P, Li Q, Xu B. Phase I Study and Biomarker Analysis of Pyrotinib, a Novel Irreversible Pan-ErbB Receptor Tyrosine Kinase Inhibitor, in Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer. J Clin Oncol. 2017 Sep 20;35(27):3105-3112. doi: 10.1200/JCO.2016.69.6179. Epub 2017 May 12. PMID 28498781
- See also: Related Info — http://dx.doi.org/10.21037/tbcr-20-25